CLINICAL TRIAL: NCT05007808
Title: Phase 2 Multicenter, Double-blind, Randomized, Parallel-Group, Vehicle-Controlled Study to Evaluate the Efficacy, Safety, and Local Tolerability of G001 in Patients With Osteoarthritis (OA) of the Knee
Brief Title: Efficacy and Safety of G001 in Patients With Osteoarthritis (OA) of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BUZZZ Pharmaceuticals Limited (Industry)
Collaborators: Veristat, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-G001-P2
Record Dates: First submitted 2021-07-22; First posted 2021-08-16 (Actual); Results first posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-03

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; knee; topical therapy; pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- G001 Topical Gel (Experimental): G001 Topical Gel, 4 grams applied to the index knee four times a day over 4 weeks.
  Interventions: Drug: G001 Topical Gel
- Vehicle Topical Gel (Placebo Comparator): Vehicle Topical Gel, 4 grams applied to the index knee four times a day over 4 weeks.
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: G001 Topical Gel — Non-steroidal anti-inflammatory drug for topical administration
  Arms: G001 Topical Gel
Drug: Vehicle — Vehicle Gel for topical administration
  Arms: Vehicle Topical Gel

SUMMARY:
Phase 2 multicenter, double-blind, randomized, parallel-group, vehicle-controlled study to evaluate the efficacy, safety, and local tolerability of G001 topical gel compared to matching Vehicle topical gel in patients with symptomatic OA of the knee.

Each patient's participation is approximately 7 weeks (~1 week screening, 4 weeks of treatment, and 2 weeks of post-treatment follow-up). Eligible patients with adequate OA pain in the index knee are randomized (1:1 allocation ratio) at the Baseline/Flare Visit 1.

Following screening, prior NSAID and/or acetaminophen use is discontinued to allow for washout and symptom flare. Patients are instructed to rate their worst daily and nightly pain in their daily diary, as well as to document all study drug applications and any rescue medication (acetaminophen) use for breakthrough pain. Acetaminophen may be used as rescue medication only, except within 12 hours prior to the Baseline Visit and within 12 hours prior to any post-baseline efficacy assessments (Weeks 2, 4, and 5). Patients are instructed to return to the clinic 3 to 7 days after the last study drug application for Flare Visit 2, and within approximately 2 weeks after the last study drug application for end-of-study evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of OA of the knee, meeting American College of Rheumatology (ACR) criteria for classification of idiopathic (primary) OA for at least 6 months prior to Screening
* Radiologic evidence of OA of the knee of grade 2 (mild) or grade 3 (moderate) according to Kellgren and Lawrence Radiographic Grading
* Worst daily pain (within 24 hours prior to Screening and Baseline) in the index knee between 4 and 8 on the 11-point pain NRS
* On stable analgesic therapy

At Baseline:

- Development of a flare of pain following washout of stable analgesic (NSAID and/or acetaminophen) therapy

Exclusion Criteria:

* Radiologic evidence of severe OA of the knee (Kellgren and Lawrence grade 4)
* Secondary OA of the index knee
* Any other arthritis, included but not limited to rheumatoid arthritis, psoriatic arthritis, etc.
* History of pseudo-gout or inflammatory flare-ups
* History of severe neurological conditions
* Any other chronic pain conditions (e.g., back pain) or disabling conditions affecting the joints
* Patients who are non-ambulatory or require the use of crutches or a walker, or started using a cane within 30 days prior to Screening
* Any history of major surgery to the index knee, minor knee surgery, or injury to the index knee within 1 year prior to Screening
* Knee arthroscopy (index knee) within 3 months prior to Screening
* Planned or candidate for knee replacement or knee reconstruction surgery
* Received intra-articular viscosupplementation/hyaluronate, joint lavage, or other invasive therapies to the index knee in the past 90 days
* Treatment with or need for any of the following: (1) oral or intramuscular corticosteroids within the past 90 days; (2) intra-articular corticosteroid injection into the index knee within the past 90 days, or into any other joint within the past 30 days; (3) current use of topical corticosteroids on the index knee
* Prior stable therapy with an opioid analgesic, or anticipated need for opioid analgesic use during the study
* Use of sedative hypnotic medication, antidepressants with known analgesic effect, antipsychotics, antiepileptics, and anti-Parkinson drugs within the past 14 days
* Regular use of medication for headaches
* Anticipated use of any oral or topical NSAID (apart from the study drug) during the study
* Known sensitivity to the study drug (or any of its ingredients), or NSAIDs, or presence of contraindications, warnings, or precautions

At Baseline:

* Worst daily pain (within the past 24 hours) in the contralateral knee assessed as >2 on the 11-point pain NRS scale
* Non-compliance with the daily diary requirement during the Screening period.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre O'Keeffe, PhD, Study Director — Buzzz Pharma
Locations (10):
- Canada (10):
  - Aggarwal and Associates Limited, Brampton
  - Medicor Research Inc., Greater Sudbury
  - Manna Research, Lévis
  - Recherche GCP Research, Montreal
  - Alpha recherche Clinique (1), Québec
  - Alpha Recherche Clinique (2), Québec
  - Centre de Recherche Saint-Louis, Québec
  - G.R.M.O. (Groupe de Recherche en Maladie Osseuses) Inc., Québec
  - Recherche Clinique Sigma Inc., Québec
  - Canadian Phase Onward Inc., Toronto

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 10 study centers in Canada. A total of 210 patients with OA of the knee were randomly assigned to double-blinded treatment in the study; of these, 105 patients received G001 and 105 patients received Vehicle.
Pre-assignment Details: Following screening, prior NSAID and/or acetaminophen use was discontinued to allow for washout (3 to 7 days) and symptom flare. Eligible patients with adequate OA pain in the index knee were randomly assigned to G001 or Vehicle in a 1:1 allocation ratio.
Period: Overall Study
Arm/Group | G001 Topical Gel | Vehicle Topical Gel
Started | 105 | 105
Completed | 99 | 100
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | G001 Topical Gel | Vehicle Topical Gel | Total
Number analyzed (Participants) | 105 | 105 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (7.89) | 65.3 (8.35) | 64.8 (8.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 61 | 125
  Male | 41 | 44 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 104 | 105 | 209
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 17 | 10 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 83 | 89 | 172
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 105 | 105 | 210
Worst daily pain (11-point NRS), Index knee [Mean (Standard Deviation); unit: Score on a scale] — 11-point Numerical Rating Scale (NRS) Scores ranging from 0 to 10, with higher scores indicating worse pain.
  Score on a scale | 6.8 (1.29) | 6.4 (1.39) | 6.6 (1.35)
Worst daily pain (11-point NRS), Contralateral knee [Mean (Standard Deviation); unit: Score on a scale] — 11-point Numerical Rating Scale (NRS) Scores ranging from 0 to 10, with higher scores indicating worse pain.
  Score on a scale | 1.1 (0.78) | 0.9 (0.81) | 1.0 (0.80)
Kellgren and Lawrence Grading [Count of Participants; unit: Participants] — Kellgren and Lawrence Radiographic Grading (0 to 4, with higher grades indicating worse OA severity):
  Grade 0: No radiographic features of osteoarthritis are present; Grade 1: Doubtful joint space narrowing (JSN) and possible osteophytic lipping; Grade 2: Presence of definite osteophytes and possible JSN on anteroposterior weight-bearing radiograph; Grade 3: Multiple osteophytes, definite JSN, sclerosis, possible bony deformity; Grade 4: Large osteophytes, marked JSN, severe sclerosis and definitely bony deformity.
  Participants
    KL Grade 2 | 46 | 53 | 99
    KL Grade 3 | 59 | 52 | 111

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in WOMAC Pain Subscale Score at Week 4/EOT
Description: Changes from Baseline in WOMAC Pain Subscale Score (5-item scale, score range 0-20, with higher scores indicating worse outcome)
Time Frame: Week 4
Population: Modified intent-to-treat (mITT) population: All randomized patients who received at least 1 dose of study drug and provided both baseline/Flare Visit 1 (FV1) and Week 4/End-of-Treatment (EOT) efficacy assessments.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | G001 Topical Gel | Vehicle Topical Gel
Number analyzed (Participants) | 103 | 104
score on a scale | -5.4 (0.32) | -5.2 (0.32)
Statistical Analysis 1: Comparison: G001 Topical Gel vs Vehicle Topical Gel; Test type: Superiority — ANCOVA model with Change from Baseline to Week 4/EOT as the outcome (dependent) variable, treatment as the independent variable, and baseline score as covariate. The p-value was derived from the t-test for the comparison of adjusted LS means between the treatment groups; p = 0.6742, t-test, 2 sided; LS Mean Difference = -0.19, 95% CI 2-sided [-1.081 to 0.701]

2. Secondary Outcome: Worst Daytime Pain Severity Scores (11-point Pain NRS), Based on Daily Diary Recordings
Description: Changes from Baseline to Week 4 in Worst Daytime Pain Severity Scores on a 0-10 scale, with higher scores indicating worse outcome
Time Frame: Week 4
Population: mITT Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | G001 Topical Gel | Vehicle Topical Gel
Number analyzed (Participants) | 103 | 104
score on a scale | -2.1 (2.01) | -2.0 (2.07)

3. Secondary Outcome: Worst Nighttime Pain Severity Score (11-point NRS), Based on Daily Diary Recordings
Description: Changes from Baseline to Week 4 in Worst Nighttime Pain Severity Scores recorded on a 0-10 scale, with higher scores indicating worse outcome
Time Frame: Week 4
Population: mITT Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | G001 Topical Gel | Vehicle Topical Gel
Number analyzed (Participants) | 103 | 103
score on a scale | -2.1 (2.01) | -1.9 (2.04)

4. Secondary Outcome: Percent Reduction From Baseline in Worst Daytime Pain
Description: Percentage of Patients Achieving ≥ 20%, ≥ 30%, and ≥ 50% Reduction from Baseline in Worst Daytime Pain at Week 4/EOT
Time Frame: Week 4
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | G001 Topical Gel | Vehicle Topical Gel
Number analyzed (Participants) | 103 | 103
Participants
  ≥ 20% Reduction from BL | 70 | 68
  ≥ 30% Reduction from BL | 58 | 53
  ≥ 50% Reduction from BL | 35 | 36

5. Secondary Outcome: Percent Reduction From Baseline in Worst Nighttime Pain
Description: Percentage of Patients Achieving ≥ 20%, ≥ 30%, and ≥ 50% Reduction from Baseline in Worst Nighttime Pain at Week 4/EOT
Time Frame: Week 4
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | G001 Topical Gel | Vehicle Topical Gel
Number analyzed (Participants) | 103 | 103
Participants
  ≥ 20% Reduction from BL | 73 | 65
  ≥ 30% Reduction from BL | 59 | 56
  ≥ 50% Reduction from BL | 36 | 35

6. Secondary Outcome: Change From Baseline in WOMAC Physical Function Subscale Score at Week 4/EOT
Description: WOMAC Physical Function Subscale (17-item, score range 0-68, with higher scores indicating worse outcome)
Time Frame: Week 4
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | G001 Topical Gel | Vehicle Topical Gel
Number analyzed (Participants) | 103 | 104
score on a scale | -12.5 (1.07) | -10.4 (1.06)

7. Secondary Outcome: Change From Baseline in WOMAC Total Score at Week 4/EOT
Description: WOMAC Osteoarthritis Index Total score (24-item, score range 0-96, with higher scores indicating worse outcome)
Time Frame: Week 4
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | G001 Topical Gel | Vehicle Topical Gel
Number analyzed (Participants) | 103 | 104
score on a scale | -19.4 (1.47) | -17.1 (1.46)

8. Secondary Outcome: Change From Baseline in WOMAC Stiffness Subscale Score at Week 4/EOT
Description: WOMAC Stiffness Subscale (2-item, range of scores 0-8, with higher scores indicating worse outcome)
Time Frame: Week 4
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | G001 Topical Gel | Vehicle Topical Gel
Number analyzed (Participants) | 103 | 104
score on a scale | -1.6 (0.14) | -1.5 (0.14)

9. Secondary Outcome: Change From Baseline in WOMAC Total and Subscale Scores at Week 2
Description: Change from Baseline to Week 2 in:
  WOMAC Osteoarthritis Index Total score (24-item, score range 0-96, with higher scores indicating worse outcome) WOMAC Pain Subscale score (5-item, score range 0-20, with higher scores indicating worse pain) WOMAC Stiffness Subscale score (2-item, score range 0-8, with higher scores indicating worse stiffness) WOMAC Physical Function Subscale score (17-item, score range 0-68, with higher scores indicating worse physical function)
Time Frame: Week 2
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | G001 Topical Gel | Vehicle Topical Gel
Number analyzed (Participants) | 103 | 104
score on a scale
  WOMAC Total score, Change from BL to Week 2 | -15.7 (1.27) | -13.2 (1.25)
  WOMAC Pain score, Change from BL to Week 2 | -4.7 (0.29) | -4.4 (0.29)
  WOMAC Stiffness score, Change from BL to Week 2 | -1.4 (0.13) | -1.0 (0.13)
  WOMAC Physical Function score, Change from BL to Week 2 | -9.5 (0.93) | -8.0 (0.91)

10. Secondary Outcome: Change From Week 4 to Week 5 in WOMAC Total and Subscale Scores
Description: Change from Week 4/EOT to Week 5/Flare Visit 2 (FV2) in:
  WOMAC Osteoarthritis Index Total score (24-item, score range 0-96, with higher scores indicating worse outcome) WOMAC Pain Subscale score (5-item, score range 0-20, with higher scores indicating worse pain) WOMAC Stiffness Subscale score (2-item, score range 0-8, with higher scores indicating worse stiffness) WOMAC Physical Function Subscale score (17-item, score range 0-68, with higher scores indicating worse physical function)
Time Frame: Week 4 to Week 5
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | G001 Topical Gel | Vehicle Topical Gel
Number analyzed (Participants) | 103 | 104
score on a scale
  WOMAC Total score, Change from Week 4/EOT to Week 5/FV2 | 3.5 (0.89) | 2.7 (0.89)
  WOMAC Pain score, Change from Week 4/EOT to Week 5/FV2 | 0.8 (0.21) | 0.7 (0.21)
  WOMAC Stiffness score, Change from Week 4/EOT to Week 5/FV2 | 0.3 (0.10) | 0.3 (0.10)
  WOMAC Physical Function score, Change from Week 4/EOT to Week 5/FV2 | 2.4 (0.65) | 1.7 (0.65)

11. Secondary Outcome: Change From Baseline in Patient Global Assessment (PGA) of Disease Activity Over Time
Description: PGA of Disease Activity (DA) was assessed on a 5-point Likert scale (0 = very good; 1 = good; 2 = fair; 3 = poor; and 4 = very poor), with higher scores indicating worse outcome.
  Change from Baseline in PGA of disease activity scores was calculated and the response was classified into 3 categories according to the following rules:
  Improved - defined as either of the following:
  * For baseline Grade ≥ 2: a reduction of ≥ 2 grades from baseline
  * For baseline Grade = 1: a change in grade from 1 to 0
  Worsened - defined as either of the following:
  * For baseline Grade ≤ 2: an increase of ≥ 2 grades from baseline
  * For baseline Grade = 3: a change in grade from 3 to 4 No Change - defined as neither Improved nor Worsened
Time Frame: Weeks 2, 4 and 5
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | G001 Topical Gel | Vehicle Topical Gel
Number analyzed (Participants) | 102 | 104
Participants
  PGA of DA, Change from BL to Week 2: number analyzed (Participants) | 99 | 102
  PGA of DA, Change from BL to Week 2: Improved | 24 | 20
  PGA of DA, Change from BL to Week 2: No change | 74 | 79
  PGA of DA, Change from BL to Week 2: Worsened | 1 | 3
  PGA of DA, Change from BL to Week 4: Improved | 38 | 28
  PGA of DA, Change from BL to Week 4: No change | 64 | 72
  PGA of DA, Change from BL to Week 4: Worsened | 0 | 4
  PGA of DA, Change from BL to Week 5: number analyzed (Participants) | 100 | 100
  PGA of DA, Change from BL to Week 5: Improved | 26 | 21
  PGA of DA, Change from BL to Week 5: No change | 73 | 75
  PGA of DA, Change from BL to Week 5: Worsened | 1 | 4

12. Secondary Outcome: Change From Baseline in Investigator Global Assessment (IGA) of Disease Activity Over Time
Description: IGA of Disease Activity (DA) was assessed on a 5-point Likert scale (0 = very good; 1 = good; 2 = fair; 3 = poor; and 4 = very poor), with higher scores indicating worse outcome.
  Change from Baseline in IGA of disease activity scores was calculated and the response was classified into 3 categories according to the following rules:
  Improved - defined as either of the following:
  * For baseline Grade ≥ 2: a reduction of ≥ 2 grades from baseline
  * For baseline Grade = 1: a change in grade from 1 to 0
  Worsened - defined as either of the following:
  * For baseline Grade ≤ 2: an increase of ≥ 2 grades from baseline
  * For baseline Grade = 3: a change in grade from 3 to 4 No Change - defined as neither Improved nor Worsened
Time Frame: Weeks 2, 4 and 5
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | G001 Topical Gel | Vehicle Topical Gel
Number analyzed (Participants) | 103 | 104
Participants
  IGA of DA, Change from BL to Week 2: number analyzed (Participants) | 99 | 102
  IGA of DA, Change from BL to Week 2: Improved | 24 | 22
  IGA of DA, Change from BL to Week 2: No Change | 74 | 77
  IGA of DA, Change from BL to Week 2: Worsened | 1 | 3
  IGA of DA, Change from BL to Week 4: Improved | 39 | 29
  IGA of DA, Change from BL to Week 4: No Change | 63 | 72
  IGA of DA, Change from BL to Week 4: Worsened | 1 | 3
  IGA of DA, Change from BL to Week 5: number analyzed (Participants) | 100 | 100
  IGA of DA, Change from BL to Week 5: Improved | 30 | 21
  IGA of DA, Change from BL to Week 5: No Change | 67 | 78
  IGA of DA, Change from BL to Week 5: Worsened | 3 | 1

13. Secondary Outcome: PGA of Overall Treatment Benefit (OTB)
Description: PGA of overall treatment benefit was completed using a 5-point Likert scale (0 = very good; 1 = good; 2 = fair; 3 = poor; and 4 = very poor) after 2 and 4 weeks of treatment, with higher scores indicating worse outcome.
Time Frame: Weeks 2 and 4
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | G001 Topical Gel | Vehicle Topical Gel
Number analyzed (Participants) | 102 | 104
Participants
  PGA of OTB at Week 2: number analyzed (Participants) | 99 | 102
  PGA of OTB at Week 2: Good or Very Good | 32 | 39
  PGA of OTB at Week 2: Fair | 49 | 47
  PGA of OTB at Week 2: Poor or Very Poor | 18 | 16
  PGA of OTB at Week 4: Good or Very Good | 50 | 46
  PGA of OTB at Week 4: Fair | 36 | 38
  PGA of OTB at Week 4: Poor or Very Poor | 16 | 20

14. Secondary Outcome: IGA of Overall Treatment Benefit (OTB)
Description: IGA of overall treatment benefit was completed using a 5-point Likert scale (0 = very good; 1 = good; 2 = fair; 3 = poor; and 4 = very poor) after 2 and 4 weeks of treatment, with higher scores indicating worse outcome.
Time Frame: Weeks 2 and 4
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | G001 Topical Gel | Vehicle Topical Gel
Number analyzed (Participants) | 103 | 104
Participants
  IGA of OTB, Week 2: number analyzed (Participants) | 99 | 102
  IGA of OTB, Week 2: Very Good or Good | 32 | 40
  IGA of OTB, Week 2: Fair | 47 | 47
  IGA of OTB, Week 2: Poor or Very Poor | 20 | 15
  IGA of OTB, Week 4: Very Good or Good | 52 | 46
  IGA of OTB, Week 4: Fair | 35 | 39
  IGA of OTB, Week 4: Poor or Very Poor | 16 | 19

15. Secondary Outcome: Rescue Medication Use
Description: Only acetaminophen was permitted as rescue medication (up to 500 mg per dose and 2000 mg/day to manage breakthrough pain). No rescue medication use was allowed within 12 hours before an efficacy assessment.
Time Frame: 5 weeks
Population: mITT Population
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | G001 Topical Gel | Vehicle Topical Gel
Number analyzed (Participants) | 103 | 104
mg/day | 71.6 (66.65) | 94.6 (123.3)

16. Other Pre Specified Outcome: Number of Participants With AEs, Study Drug-related AEs, Serious AEs, and AEs Leading to Study Drug Discontinuation
Description: Number and percentage of participants with adverse events (AEs), study drug-related AEs, serious AEs, and AEs leading to study drug discontinuation
Time Frame: 6 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | G001 Topical Gel | Vehicle Topical Gel
Number analyzed (Participants) | 105 | 105
Participants
  Any TEAE | 36 | 28
  Treatment-related TEAEs | 5 | 4
  Any SAE | 0 | 1
  Any TEAE leading to Discontinuation | 3 | 1

17. Other Pre Specified Outcome: Frequency and Severity of Application Site AEs
Description: Number and percentage of participants with application site AEs
Time Frame: 6 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | G001 Topical Gel | Vehicle Topical Gel
Number analyzed (Participants) | 105 | 105
Participants | 0 | 1

18. Other Pre Specified Outcome: Skin Irritation Test Scores (Berger/Bowman Scoring Scale)
Description: The Numerical Total Score is the sum of the Dermal Response score (from 0=No evidence of irritation to 7=Strong reaction spreading beyond the application site) and the numeric equivalent of Other Effects score (from 0=Slightly glazed appearance to 3=Small petechial erosions and/or scabs).
  The Numerical Total Score range is from 0 to 10, with higher scores indicating worse outcome/skin irritation.
Time Frame: Weeks 2, 4, and 6
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | G001 Topical Gel | Vehicle Topical Gel
Number analyzed (Participants) | 103 | 104
Participants
  Skin Irritation Total Score, Week 2: number analyzed (Participants) | 100 | 102
  Skin Irritation Total Score, Week 2: Numerical Total Score of 0 | 98 | 101
  Skin Irritation Total Score, Week 2: Numerical Total Score of 1 | 1 | 0
  Skin Irritation Total Score, Week 2: Numerical Total Score of ≥2 | 1 | 1
  Skin Irritation Total Score, Week 4/EOT: Numerical Total Score of 0 | 101 | 103
  Skin Irritation Total Score, Week 4/EOT: Numerical Total Score of 1 | 1 | 1
  Skin Irritation Total Score, Week 4/EOT: Numerical Total Score of ≥2 | 1 | 0
  Skin Irritation Total Score, Week 6: number analyzed (Participants) | 101 | 101
  Skin Irritation Total Score, Week 6: Numerical Total Score of 0 | 101 | 101
  Skin Irritation Total Score, Week 6: Numerical Total Score of 1 | 0 | 0
  Skin Irritation Total Score, Week 6: Numerical Total Score of ≥2 | 0 | 0

19. Other Pre Specified Outcome: ECG Abnormalities in QT, QTc, QRS, or PR Intervals
Description: Number and percentage of participants with clinically significant (CS) abnormal results in QT, QTc, QRS, or PR intervals at Week 4/EOT
Time Frame: 4 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | G001 Topical Gel | Vehicle Topical Gel
Number analyzed (Participants) | 105 | 105
Participants
  CS QT Interval abnormality | 0 | 0
  CS QTc Interval abnormality | 0 | 0
  CS QRS Interval abnormality | 0 | 0
  CS PR Interval abnormality | 0 | 0

20. Other Pre Specified Outcome: Changes From Baseline in Safety Laboratory Test Results
Description: Mean changes (descriptive) and shifts from normal baseline to laboratory values outside reference ranges
Time Frame: 6 weeks
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Changes in Vital Signs Measurements
Description: Mean changes (descriptive) from baseline
Time Frame: 6 weeks
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Changes in Physical Examination
Description: Number and percentage of participants with clinically significant abnormal findings
Time Frame: 6 weeks
Reporting Status: Not Posted

23. Secondary Outcome: Number of Rescue Medication Doses
Description: as for outcome 15
Time Frame: 5 weeks
Population: mITT Population
Measure: Mean (Standard Deviation); unit: number of doses
Arm/Group | G001 Topical Gel | Vehicle Topical Gel
Number analyzed (Participants) | 103 | 104
number of doses | 5.9 (6.03) | 7.9 (12.54)

ADVERSE EVENTS:
Time Frame: Adverse event (AE) collection period: from the Screening Visit (Day -7 to -3) to the Week 6/End-of-Study (EOS) Visit (Day 43 +/-3). Analyses of AEs were performed for treatment-emergent events (TEAEs), defined as any AE with onset during or after the first application of study drug through the end of the study (Week 6/EOS visit), or any event that was present at Baseline but worsened in severity during or after the first application of study drug.
Description: Adverse events of special interest for G001 included application site adverse reactions.
  All AEs occurring between the Screening visit and the Week 6/EOS visit were recorded in the patient's medical record and eCRF.
Arm/Group | G001 Topical Gel | Vehicle Topical Gel
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/105 | 1/105
Other Adverse Events (participants affected / at risk) | 10/105 | 5/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G001 Topical Gel (N=105) | Vehicle Topical Gel (N=105)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) — Reported Term: Tachycardic atrial fibrillation Assessed as moderate in intensity, and not related to the (blinded) study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G001 Topical Gel (N=105) | Vehicle Topical Gel (N=105)
Headache (Nervous system disorders) | 10 (14) | 5 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/08/NCT05007808/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/08/NCT05007808/SAP_001.pdf